CLINICAL TRIAL: NCT01526746
Title: An Open-Label, Single-Dose, Parallel-Group Study to Compare the Pharmacokinetics of Tasimelteon in Subjects With Renal Impairment With That in Matched Control Subjects With Relatively Normal Renal Function
Brief Title: Pharmacokinetics of Tasimelteon in Subjects With Renal Impairment and Matched Control Subjects With Relatively Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VP-VEC-162-1106
Record Dates: First submitted 2012-01-26; First posted 2012-02-06 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Renal Impairment
Keywords: End stage renal disease; ESRD; kidney disease; renal impairment; renal
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic; Kidney Diseases | interventions — tasimelteon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- End Stage Renal Disease, dialysis (Experimental): eGFR <15 ml/min/1.73m^2
  Interventions: Drug: Tasimelteon
- Severe renal impairment (Experimental): eGFR < 29 ml/min/1.73m^2
  Interventions: Drug: Tasimelteon
- Healthy controls (Experimental): eGFR > 80 mL/min/1.73m^2 Matched to renally impaired subjects by age, gender, BMI, and smoking status
  Interventions: Drug: Tasimelteon

INTERVENTIONS:
Drug: Tasimelteon — 20mg capsule, once
  Other Names: VEC-162
Drug: Tasimelteon — 20mg, once

SUMMARY:
The purpose of this research study is to understand whether there is any difference in the amount of tasimelteon (including its breakdown products) in the blood of individuals with severe renal impairment compared to individuals who have normal renal function. The safety and tolerability of tasimelteon will also be assessed throughout this study.

ELIGIBILITY:
Inclusion Criteria:

Groups 1-3

1. Ability and acceptance to provide written informed consent;
2. Men or women between 18 - 79 years, inclusive;
3. Subjects with Body Mass Index (BMI) of >18 and <40 kg/m2 (BMI = weight (kg)/ [height (m)]2);
4. Males, non-fecund females (i.e., surgically sterilized, if procedure was done 6 months before screening or subject is postmenopausal, without menses for 6 months before screening), or females of child-bearing potential using an acceptable method of birth control for a period of 35 days before the first dosing and have a negative pregnancy test at the screening and baseline visits; Note 1: Acceptable methods of birth control include any one of the following: abstinence, vasectomized sexual partner, hormonal methods (i.e. pill, hormonal IUD, Depo-Provera, implants, patch, intravaginal device [NuvaRing]), intrauterine device (IUD [copper banded coils]), diaphragm, cervical cap, or condom with spermicidal jelly or foam.
5. Willing and able to comply with study requirements and restrictions;

Groups 1- 2 (renal impairment)

1. Subjects with renal impairment defined as

   1. Group 1: Stage 5 End Stage Renal Disease (ESRD) (eGFR < 15 mL/min/m2) requiring regularly scheduled dialysis and have been on a stable dialysis regimen for at least three months at baseline; OR
   2. Group 2: Stage 4 severe renal impairment (eGFR ≤ 29 mL/min/m2) but not requiring dialysis as calculated using the Modification of Diet in Renal Disease (MDRD) Equation (Appendix 18.3)
2. Otherwise considered healthy in general as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening;
3. Vital signs (after 3 minutes resting in a semi-supine position) which are within the ranges shown below.

   1. Body temperature between 35.0-37.5 °C;
   2. Systolic blood pressure between 100-180 mmHg;
   3. Diastolic blood pressure between 60-115 mmHg;
   4. Pulse rate between 40-100 bpm.

Group 3 (healthy matched controls)

1. Subjects in Group 3 must match in gender, smoking status, age (±10 years), and body mass index [normal BMIs (18.00-24.99), overweight BMIs (25.00-30.99) and obese BMIs (31.00-40.00)] to Group 1 and/or 2;
2. Subjects must have normal renal function defined as eGFR ≥ 80 mL/min/m2 as calculated using the Modification of Diet in Renal Disease (MDRD) Equation (Appendix 18.3 );
3. Subjects must be in good health as determined by past medical history, physical examination, electrocardiogram, laboratory tests and urinalysis;
4. Vital signs (after 3 minutes resting in a semi-supine position) which are within the ranges shown below:

   1. Body temperature between 35.0 - 37.5 °C;
   2. Systolic blood pressure between 90 - 150 mmHg;
   3. Diastolic blood pressure between 50 - 95 mmHg;
   4. Pulse rate between 40 - 90 bpm.

Exclusion Criteria:

Groups 1-3

1. Smokers (use of tobacco products in the previous 3 months) unable or unwilling to limit consumption to 10 cigarettes per day or less while checked into the inpatient facility.

   a. Note: Smoking will be a match criteria and the site should attempt to enroll an equal number of smokers and non-smokers into each group.
2. Exposure to any investigation drug, including placebo, within 30 days or 5 half-lives (whichever is longer) of dosing;
3. Donation or loss of 400 mL or more of blood within two months prior to dosing;
4. Significant illness within the two weeks prior to dosing;
5. Answer 'yes' to either Question 4 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan) or Question 5 (Active Suicidal Ideation with Specific Plan and Intent) on the "Suicidal Ideation" portion of the C-SSRS, or answer "yes" to any of the suicide-related behaviors (actual attempt, interrupted attempt, aborted attempt, preparatory act, or behavior) on the "Suicidal Behavior" portion of the Columbia Suicide Severity Rating Scale (C-SSRS); and the ideation or behavior occurred within the past 6 months;
6. Functioning renal transplant;
7. History within the past 2 years of clinically significant acute or chronic bronchospastic disease, including asthma and chronic obstructive pulmonary disease, treated or not treated;
8. Treatment with any drug known to cause major organ system toxicity (e.g., chloramphenicol or tamoxifen) during the 60 day preceding the Screening visit;
9. Participation in a previous BMS-214778/VEC-162 trial;
10. History of drug or alcohol abuse as defined in DSM-IV, Diagnostic Criteria for Drug and Alcohol Abuse, within the 12 months prior to screening or evidence of such abuse as indicated by the laboratory assays conducted during the screening and baseline visits. A positive drug screen in Groups 1 and 2 is acceptable if there is documentation that subjects have been prescribed the corresponding medication;
11. History of immunocompromise, including a positive HIV (ELISA and Western blot) test result;
12. A positive Hepatitis B surface antigen (HBsAg) test result;
13. Any surgical or medical condition which might significantly alter the absorption, distribution or excretion of any drug. The Investigator should be guided by evidence of any of the following:

    1. History of clinically significant inflammatory bowel syndrome, gastritis, ulcers, gastrointestinal or rectal bleeding;
    2. History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection;
    3. History of pancreatic injury or pancreatitis;
    4. History or presence of liver disease or liver injury as indicated by lab values such as SGOT, SGPT, GGT, alkaline phosphatase, or serum bilirubin 1.5 times greater than the upper limit of normal;
14. Clinically significant ECG abnormalities or vital sign abnormalities at screening or a history of unstable, severe, or clinically significant cardiovascular disease (e.g., myocardial infarction within previous 6 months, unstable angina, cardiac failure, second/third degree atrioventricular block);
15. Subjects taking any unapproved prescription or over-the-counter medications; all concomitant medications must be discussed with and approved by the sponsor prior to enrollment;
16. A known hypersensitivity to tasimelteon or drugs similar to tasimelteon including melatonin;
17. Pregnant or lactating females;
18. Inability to swallow the study medication whole;
19. Any other sound medical reason as determined by the clinical Investigator.

Groups 1 - 2 (renal impairment)

1. Subjects with clinically significant abnormal findings, not consistent with clinical disease, upon physical examination, ECG, or laboratory evaluation;
2. Evidence of progressive renal disease within 4 weeks prior to screening;
3. Acute renal failure or nephrotic syndrome;
4. Current hematuria of urologic origin;
5. Any significant change in chronic treatment medication as determined by the clinical Investigator.

Group 3 (healthy matched controls)

1. Use of unapproved prescription medication within 1 month of dosing and OTC medication within 14 days prior to dosing;
2. History or presence of impaired renal function as indicated by abnormal (>ULN) creatinine or BUN values or abnormal urinary constituents (e.g., albuminuria).
3. A positive hepatitis C test result.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Tasimelteon pharmacokinetic parameters (AUC, Cmax, Tmax) | Predose, 0.25, 1, 1.5, 2, 4, 6, 8, 12, 24, 30, and 36 hours post-dose

SECONDARY OUTCOMES:
Pharmacokinetic parameters (AUC, Cmax, Tmax) of tasimelteon metabolites M3, M9, M11, M12, M13, and M14 | Predose, 0.25, 1, 1.5, 2, 4, 6, 8, 12, 24, 30, and 36 hours post-dose
The percentage of tasimelteon and its metabolites that are removed by hemodialysis (AUC) | 4, 6, 8 hours after dosing
  paired arterial and venous samples
The ratio of plasma protein bound versus unbound fractions of tasimelteon and metabolites M9, M11, M12, M13, and M14 | 0.5 and 3 hours post dose
Safety and tolerability as measured by spontaneous reporting of AEs, and clinically significant changes in laboratory parameters, ECG parameters, and vital signs | 36 hours
The Columbia-Suicide Severity Rating Scale will be used to assess suicidal behavior and ideation. | once per day at Screening (approximately day -7), Day -1 (baseline), Day 2 (end of study)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Clinical Pharmacology of Miami, Inc., Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - DaVita Clinical Research, Minneapolis, Minnesota